CLINICAL TRIAL: NCT05701774
Title: An Open-Label Study of DCCR (Diazoxide Choline) Extended-Release Tablets in Patients With Prader-Willi Syndrome
Brief Title: Open-Label Extension Study of DCCR in Patients With Prader-Willi Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Soleno Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C614
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DCCR (Experimental): 75 - 525 mg DCCR
  Interventions: Drug: DCCR

INTERVENTIONS:
Drug: DCCR — Once daily oral administration

SUMMARY:
The purpose of this is study is to evaluate the long-term safety of DCCR (diazoxide choline) extended-release tablets) in patients with Prader-Willi syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Provide voluntary, written informed consent (parent(s) / legal guardian(s) of patient); provide voluntary, written assent (subjects, as appropriate)
2. Participant must:

   1. Have participated in and completed the Study C602 Randomized Withdrawal (RW) Period;
   2. Have participated in but discontinued from the Study C602 RW Period and at least 16 weeks have elapsed since the date of their randomization into the C602 RW Period; or
   3. Have participated in Study C602 OLE period, did not consent to participate in the RW Period, and at least 16 weeks have elapsed since the date of their C602 Open-Label Extension End of Treatment Visit.

Exclusion Criteria:

1. Positive urine pregnancy test (in females of child-bearing potential)
2. Females who are pregnant or breastfeeding, and/or plan to become pregnant or to breast-feed during or within 30 days after study participation.
3. Participation in a clinical study of an investigational drug (including approved drugs for unapproved uses), investigational device, or therapeutic intervention subsequent to the C602 Open-Label Extension End of Treatment Visit.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Safety of DCCR (adverse events. Safety analyses will be conducted in all subjects who receive at least one dose of DCCR in the C614 study. ( Adverse events) | Baseline to End of Study or until resolution of certain adverse events
  Assess the safety of DCCR by evaluating the incidence and severity of adverse events.
  Safety analyses will be conducted in all subjects who receive at least one dose of DCCR in the C614 study. Adverse events will be described by type and level of severity.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (17):
  - UC Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital of San Diego, San Diego, California
  - U of Florida Gainesville, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - National Institutes of Health, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Children's Hospital and Clinic Minnesota, Saint Paul, Minnesota
  - St. Joseph's University Medical Center, Paterson, New Jersey
  - NYU Winthrop Hospital, Mineola, New York
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's, Seattle, Washington
- United Kingdom (5):
  - Fulbourn Hospital, Cambridge
  - The Queen Elizabeth University, Glasgow
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Royal London Hospital, London
  - Chelsea and Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No